CLINICAL TRIAL: NCT05074745
Title: Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Buccal Screening Evaluation Using an RT-PCR Assay and a Rapid ELISA Test Among Symptomatic and Asymptomatic Patients: the CORDAGES Study
Brief Title: Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Buccal Screening Evaluation Using an RT-PCR Assay and a Rapid ELISA Test Among Symptomatic and Asymptomatic Patients
Acronym: CORDAGES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Scientifique de Monaco (Other)
Collaborators: Department of Health Affairs, Monaco (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO_CSM_01_2021
Record Dates: First submitted 2021-10-07; First posted 2021-10-12 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: SARS-CoV-2; COVID-19
Keywords: SARS-CoV-2; POCT; RT-PCR; Contact case; ELISA; Buccal
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Monocentric, Prospective, 3 components Nasopharyngeal swab by PCR Buccal swab by PCR Buccal by ELISA POCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Buccal and nasopharyngeal swabs (Experimental): One patient will have 3 swabs taken, 2 buccal for PCR and ELISA POCT, 1 nasopharyngeal for PCR
  Interventions: Diagnostic Test: ELISA POCT vs RT-PCR

INTERVENTIONS:
Diagnostic Test: ELISA POCT vs RT-PCR — 3 swabs taken, buccal for RT-PCR and ELISA POCT, nasopharyngeal for RT-PCR

SUMMARY:
The main objective is to expand screening for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) by evaluating the diagnostic accuracy of the RT-PCR test (Cobas® Roche, Switzerland) and the ELISA Point of Contact Testing (PORTABLE COVID-19 ANTIGEN LAB® Stark, Italy) on buccal swab compared to the reference test, the RT-PCR test (Cobas® Roche, Switzerland) on nasopharyngeal swab.

Secondary objectives

* To evaluate the diagnostic accuracy of oral swab RT-PCR and POCT relative to the quantitative amplification (Ct) values of the NP Swab RT-PCR assay.
* Analyze RT-PCR amplification cycle thresholds (Ct) and POCT diagnostic accuracy as a function of the presence and timing of symptoms.
* Among symptomatic participants, compare clinical presentations between positive and negative participants on the NP swab RT-PCR test.
* The RT-PCR test may be imperfectly sensitive, ranging from 71 to 98%3. Using a Bayesian latent class model, the investigators will assess the true accuracy of POCT as it does not require the assumption that any one test or combination of tests is perfect14,15.

ELIGIBILITY:
Inclusion Criteria:

* 18+ patient eligible for COVID-19 testing in Monaco
* symptoms suggestive of COVID-19
* contact with a confirmed case of COVID-19

Exclusion Criteria:

* refusal to participate in the study
* preventive screening of professional groups
* inability to return to the screening center within 48-72 hours of the first visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2021-02-18 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) positive patients for the two different sampling types (buccal vs nasopharyngeal) and two methods (ELISA POCT vs RT-PCR) | 48 Hours
  Number of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) positive patients by sampling type (buccal and nasopharyngeal swab) and analytical method (ELISA POCT vs RT-PC)

SECONDARY OUTCOMES:
Comparison of Ct values in buccal and nasopharyngeal swabs | 48 Hours
  Ct values by PCR in buccal and nasopharyngeal swabs

CONTACTS AND LOCATIONS:
Locations (1):
- Centre National de Depistage - Espace Leo Ferre, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Althaus T, Blake A, Costantini A, Lavagna C, Jacquesson E, Groshenry G, Troel A, Vanzo B, Dejoux O, Raps H, Rampal P, Voiglio EJ. Diagnostic accuracy of non-invasive SARS-CoV-2 screening tests: a national prospective analysis. BMC Infect Dis. 2025 May 21;25(1):727. doi: 10.1186/s12879-025-11088-x. PMID 40399889